CLINICAL TRIAL: NCT02229851
Title: A Multicentre, Multinational, Randomised, Parallel-group, Placebo-controlled (Double Blind) and Active-controlled (Open) Trial to Compare the Efficacy and Safety of Once Weekly Dosing of NNC0195-0092 (Somapacitan) With Once Weekly Dosing of Placebo and Daily Norditropin® FlexPro® in Adults With Growth Hormone Deficiency for 35 Weeks, Followed by a 53-week Open-label Extension Period
Brief Title: Trial to Compare the Efficacy and Safety of NNC0195-0092 (Somapacitan) With Placebo and Norditropin® FlexPro® (Somatropin) in Adults With Growth Hormone Deficiency.
Acronym: REAL 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8640-4054; 2013-002892-16 (Registry Identifier: European Medicines Agency); U1111-1145-0211 (Other: World Health Organization (WHO)); JapicCTI-152767 (Registry Identifier: JAPIC)
Record Dates: First submitted 2014-08-26; First posted 2014-09-03 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan; NNC0195-0092; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NNC0195-0092 (somapacitan) (Experimental)
  Interventions: Drug: somapacitan
- Daily hGH (Active Comparator)
  Interventions: Drug: somatropin
- Placebo (Placebo Comparator): Switch to NNC0195-0092 (somapacitan) treatment in the extension period.
  Interventions: Drug: somapacitan; Drug: placebo

INTERVENTIONS:
Drug: somapacitan — Administered subcutaneously (s.c., under the skin) once weekly for 26 weeks following 8 weeks of titration. Extension of 44 weeks' treatment following 8 weeks of titration.
  Other Names: NNC0195-0092
  Arms: NNC0195-0092 (somapacitan); Placebo
Drug: somatropin — Administered subcutaneously (s.c., under the skin) once daily for 26 weeks following 8 weeks of titration. Re-randomisation to extension of 44 weeks' treatment following 8 weeks of titration.
  Arms: Daily hGH
Drug: placebo — Administered subcutaneously (s.c., under the skin) once weekly for 26 weeks following 8 weeks of titration.
  Arms: Placebo

SUMMARY:
This study is conducted globally. The purpose is to demonstrate the efficacy of once weekly dosing of NNC0195-0092 (somapacitan) compared to placebo and once-daily dosing of somatropin (human growth hormone, hGH) after 35 weeks of treatment in adults with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 23 years of age and not more than 79 years of age at the time of signing informed consent
* Human growth hormone (hGH) treatment naïve or no exposure to hGH or growth hormone (GH) secretagogues for at least 180 days prior to randomisation with any registered or investigational hGH or GH secretagogue product (if only used in connection with stimulation tests for diagnosis of growth hormone deficiency (GHD), subjects can be included)
* If applicable, hormone replacement therapies for any other hormone deficiencies, adequate and stable for at least 90 days prior to randomisation as judged by the investigator
* FOR ALL COUNTRIES EXCEPT JAPAN:

Confirmed diagnosis of adult growth hormone deficiency (Subjects must satisfy one of the following criterion and documentation of test results must be available before randomisation (either from subjects' file or new test):

1. Insulin tolerance test (ITT) or glucagon test: a peak GH response of less than 3 ng/mL (3 mcg/L)
2. Growth hormone releasing hormone (GHRH) + arginine test according to body mass index (BMI): i) BMI less than 25 kg/m^2, a peak GH less than 11 ng/mL (11 mcg/L), ii) BMI 25-30 kg/m^2, a peak GH less than 8 ng/mL (8 mcg/L), iii) BMI greater than 30 kg/m^2, a peak GH less than 4 ng/mL (4 mcg/L)
3. Three or more pituitary hormone deficiencies and insulin like growth factor - I standard deviation score (IGF-I SDS) less than -2.0 - FOR JAPAN ONLY: Confirmed diagnosis of adult growth hormone deficiency (subjects with adult onset adult growth hormone deficiency (AGHD) need to satisfy at least one of the following criteria, subjects with a history of childhood GHD need to satisfy at least 2 of the following criteria):

a. ITT test: a peak GH of less than or equal to 1.8 ng/mL (assay using recombinant GH standard) b. glucagon test: a peak GH of less than or equal to 1.8 ng/mL (assay using recombinant GH standard) c. growth hormone releasing peptide 2 (GHRP-2) tolerance test: a peak GH of less than or equal to 9 ng/mL (assay using recombinant GH standard)

Exclusion Criteria:

* Active malignant disease or history of malignancy. Exceptions to this exclusion criterion: - Resection in situ carcinoma of the cervix uteri. Complete eradication of squamous cell or basal cell carcinoma of the skin
* Subjects with GHD attributed to treatment of intracranial malignant tumours or leukaemia, provided that a recurrence-free survival period of at least 5 years is documented in the subject's file

Ages: 23 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure' (1452), Study Director — Novo Nordisk A/S
Locations (107):
- United States (26):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Reno, Nevada
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Shavano Park, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Federal Way, Washington
  - Novo Nordisk Investigational Site, Seattle, Washington
- Australia (8):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
  - Novo Nordisk Investigational Site, Darlinghurst, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Woolloongabba, Queensland
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Nedlands, Western Australia
- Novo Nordisk Investigational Site, São Paulo, São Paulo, Brazil
- Germany (4):
  - Novo Nordisk Investigational Site, Aachen
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Oldenburg
- India (8):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Hyderabad, Telangana
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Israel (3):
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Japan (15):
  - Novo Nordisk Investigational Site, Bunkyo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Hamamatsu-shi, Shizuoka
  - Novo Nordisk Investigational Site, Itabashi-ku, Tokyo
  - Novo Nordisk Investigational Site, Kagoshima
  - Novo Nordisk Investigational Site, Kyoto-shi Kyoto
  - Novo Nordisk Investigational Site, Minato-ku, Tokyo
  - Novo Nordisk Investigational Site, Okayama, Okayama
  - Novo Nordisk Investigational Site, Sagamihara-shi, Kanagawa
  - Novo Nordisk Investigational Site, Sapporo, Hokkaido
  - Novo Nordisk Investigational Site, Sappro-shi, Hokkaido
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yamagata-shi, Yamagata
  - Novo Nordisk Investigational Site, Yokohama, Kanagawa
- Novo Nordisk Investigational Site, Riga, Latvia
- Lithuania (2):
  - Novo Nordisk Investigational Site, Kaunas
  - Novo Nordisk Investigational Site, Vilnius
- Malaysia (3):
  - Novo Nordisk Investigational Site, Kuching
  - Novo Nordisk Investigational Site, Pulau Pinang
  - Novo Nordisk Investigational Site, Putrajaya
- Novo Nordisk Investigational Site, Oslo, Norway
- Poland (5):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Romania (6):
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Iași
  - Novo Nordisk Investigational Site, Sibiu
  - Novo Nordisk Investigational Site, Timișoara
- Russia (5):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Krasnoyarsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Tomsk
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Tygerberg, Western Cape
- Sweden (3):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Uppsala
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Kocaeli
- Ukraine (2):
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Kyiv
- United Kingdom (7):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Johannsson G, Gordon MB, Hojby Rasmussen M, Hakonsson IH, Karges W, Svaerke C, Tahara S, Takano K, Biller BMK. Once-weekly Somapacitan is Effective and Well Tolerated in Adults with GH Deficiency: A Randomized Phase 3 Trial. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1358-76. doi: 10.1210/clinem/dgaa049. PMID 32022863
- [Derived] Otsuka F, Rasmussen MH, Endo T, Svaerke C, Tahara S, Johannsson G. Efficacy in Japanese adults with growth hormone deficiency receiving weekly somapacitan or daily growth hormone: results from phase 3 REAL 1 trial. Front Endocrinol (Lausanne). 2025 Feb 7;16:1534891. doi: 10.3389/fendo.2025.1534891. eCollection 2025. PMID 39991735
- [Derived] Takahashi Y, Biller BMK, Fukuoka H, Ho KKY, Rasmussen MH, Nedjatian N, Svaerke C, Yuen KCJ, Johannsson G. Weekly somapacitan had no adverse effects on glucose metabolism in adults with growth hormone deficiency. Pituitary. 2023 Feb;26(1):57-72. doi: 10.1007/s11102-022-01283-3. Epub 2022 Nov 15. PMID 36380045
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 92 sites in 16 countries: Australia - 8, Germany - 4, India - 5, Japan - 14, Latvia - 1, Lithuania - 2, Malaysia - 3, Poland - 5, Romania - 5, Russian Fed. - 6, South Africa - 3, Sweden - 1, Turkey - 4, Ukraine - 1, United Kingdom - 4, United States - 26.
Pre-assignment Details: The trial had a main phase and an extension phase. Participants were treated for 34 weeks in the main phase (followed by 1 week washout) and for 52 weeks in the extension phase (followed by 1 week washout).300 participants received treatment;1 participant was randomised but didn't receive any treatment and was therefore not included in any analyses
Groups:
- Placebo: Participants received placebo matched to somapacitan for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
- Norditropin: Participants recieved Norditropin® FlexPro® 10 mg/1.5 mL for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
- Somapacitan: Participants received Somapacitan PDS290 10mg/1.5mL for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
- Placebo/Somapacitan: Participants who received placebo in the main period, were switched to receive somapacitan for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
- Somapacitan/Somapacitan: Participants who received somapacitan in the main period, continued to receive somapacitan for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
- Norditropin/Norditropin: Participants who received Norditropin in the main phase were randomised 1:1 to continue with norditropin or switch to somapacitan. Participants who received Norditropin in the main period, continued to receive Norditropin for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
- Norditropin/Somapacitan: Participants who received Norditropin in the main phase were randomised 1:1 to continue with Norditropin or switch to somapacitan. Participants who received Norditropin in the main period, were switched to receive somapacitan for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
Period: Main Phase (Double-blind Phase)
Arm/Group | Placebo | Norditropin | Somapacitan | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Started | 61 | 119 | 120 | 0 (This arm is not applicable for the Main phase.) | 0 (This arm is not applicable for the Main phase.) | 0 (This arm is not applicable for the Main phase.) | 0 (This arm is not applicable for the Main phase.)
Full Analysis Set | 61 | 119 | 120 | 0 | 0 | 0 | 0
Safety Analysis Set | 61 | 119 | 120 | 0 | 0 | 0 | 0
Completed | 55 | 103 | 114 | 0 | 0 | 0 | 0
Not Completed | 6 | 16 | 6 | 0 | 0 | 0 | 0
Not completed — Unclassified | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 12 | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase (Open-label Phase)
Arm/Group | Placebo | Norditropin | Somapacitan | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Started | 0 (This arm is not applicable for the Extension phase.) | 0 (This arm is not applicable for the Extension phase.) | 0 (This arm is not applicable for the Extension phase.) | 55 | 114 | 52 | 51
Completed | 0 | 0 | 0 | 53 | 109 | 47 | 48
Not Completed | 0 | 0 | 0 | 2 | 5 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4 | 3 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Norditropin: Participants received Norditropin® FlexPro® 10 mg/1.5 mL for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
  Participants were re-randomised to receive somapacitan while other continued to receive Norditropin for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension part of the trial.
- Somapacitan: Participants received Somapacitan PDS290 10mg/1.5mL for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial. Participants continued to receive somapacitan for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
- Total: Total of all reporting groups
Arm/Group | Placebo | Norditropin | Somapacitan | Total
Number analyzed (Participants) | 61 | 119 | 120 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (15.7) | 45.7 (15.3) | 44.6 (14.3) | 45.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 61 | 62 | 155
  Male | 29 | 58 | 58 | 145
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Asian | 16 | 36 | 34 | 86
    Black or African American | 2 | 3 | 2 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    White | 42 | 76 | 82 | 200
    Other: Hispanic | 1 | 0 | 1 | 2
    Other: Hispanic or Latino | 0 | 1 | 0 | 1
    Other: Caucasian | 0 | 1 | 0 | 1
    Not applicable | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 4 | 8 | 6 | 18
    Not Hispanic or Latino | 57 | 109 | 114 | 280
    Not applicable | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Truncal Fat Percentage (Week 34)
Description: Change in Truncal fat percentage was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of truncal fat
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 111 | 116
Percentage of truncal fat | 0.49 (3.31) | -2.39 (4.48) | -1.17 (2.89)
Statistical Analysis 1: Comparison: Placebo vs Somapacitan; Changes in truncal fat percentage from baseline to the 34 week's measurements was analysed using an analysis of covariance model with treatment, growth hormone deficiency (GHD) onset type, sex, region, diabetes mellitus (DM) and sex by region by DM interaction as factors and baseline as a covariate. The analysis was conducted using a multiple imputation technique where trajectory after a withdrawn subjects last observation was imputed based on data from the placebo arm; Test type: Superiority; p = 0.0090, ANCOVA; Treatment difference = -1.53, 95% CI 2-sided [-2.68 to -0.38] — Somapacitan-Placebo

2. Secondary Outcome: Change in Truncal Fat Percentage (Week 87)
Description: Change in Truncal fat percentage was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of truncal fat
Groups:
- Norditropin/Norditropin: Participants who received Norditropin in the main period, continued to receive Norditropin for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
- Norditropin/Somapacitan: Participants who received Norditropin in the main period, were switched to receive somapacitan for 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment) in the extension period of the trial.
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 52 | 109 | 48 | 47
Percentage of truncal fat | -2.16 (3.94) | -1.63 (3.65) | -2.63 (4.65) | -0.96 (4.51)

3. Secondary Outcome: Change in Truncal Fat Mass (Week 34)
Description: Change in Truncal fat mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 111 | 116
grams | 417.86 (1536.36) | -619.67 (1887.50) | -180.98 (1762.31)

4. Secondary Outcome: Change in Truncal Fat Mass (Week 87)
Description: Change in Truncal fat mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 52 | 109 | 48 | 47
grams | -311.85 (1771.78) | -196.18 (2249.21) | -685.56 (2258.93) | 364.08 (2548.85)

5. Secondary Outcome: Change in Truncal Lean Body Mass (Week 34)
Description: Change in Truncal lean body mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 111 | 116
grams | 402.69 (1247.67) | 832.77 (1409.74) | 800.27 (1377.75)

6. Secondary Outcome: Change in Truncal Lean Body Mass (Week 87)
Description: Change in Truncal lean body mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 52 | 109 | 48 | 47
grams | 1197.30 (1500.56) | 1152.79 (1480.06) | 975.79 (1258.62) | 1015.12 (1554.88)

7. Secondary Outcome: Change in Total Fat Mass (Week 34)
Description: Change in Total fat mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 111 | 116
grams | 305.47 (2689.06) | -855.71 (3167.06) | -85.47 (3022.71)

8. Secondary Outcome: Change in Total Fat Mass (Week 87)
Description: Change in total fat mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: Week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 52 | 109 | 48 | 47
grams | -540.04 (3250.16) | -118.07 (3795.36) | -923.01 (4099.45) | 874.56 (4789.34)

9. Secondary Outcome: Change in Visceral Adipose Tissue (Week 34)
Description: Change in Visceral adipose tissue was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: centimeter square
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 53 | 104 | 105
centimeter square | 4.41 (13.81) | -9.68 (21.37) | -11.61 (23.93)

10. Secondary Outcome: Change in Visceral Adipose Tissue (Week 87)
Description: Change in Visceral adipose tissue was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: Week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: centimeter square
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 48 | 97 | 40 | 43
centimeter square | -9.34 (25.67) | -6.71 (33.07) | -5.17 (20.11) | -5.97 (28.86)

11. Secondary Outcome: Change in Android Fat Mass (Week 34)
Description: Change in Android fat mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 55 | 110 | 114
gram | 56.32 (293.93) | -158.98 (325.35) | -81.52 (361.62)

12. Secondary Outcome: Change in Android Fat Mass (Week 87)
Description: Change in Android fat mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 51 | 107 | 47 | 47
gram | -107.16 (367.14) | -39.76 (481.66) | -100.76 (386.24) | 11.52 (489.85)

13. Secondary Outcome: Change in Gynoid Fat Mass (Week 34)
Description: Change in Gynoid fat mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 55 | 110 | 114
gram | 8.35 (567.04) | -128.59 (471.00) | 22.66 (510.45)

14. Secondary Outcome: Change in Gynoid Fat Mass (Week 87)
Description: Change in Gynoid fat mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 51 | 107 | 47 | 47
gram | -92.00 (759.37) | 10.23 (557.20) | -100.97 (620.16) | 140.02 (790.74)

15. Secondary Outcome: Change in Appendicular Skeletal Muscle Mass (Week 34)
Description: Change in Appendicular skeletal muscle mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 111 | 116
gram | -76.22 (1006.58) | 482.76 (1246.89) | 565.21 (1011.18)

16. Secondary Outcome: Change in Appendicular Skeletal Muscle Mass (Week 87)
Description: Change in Appendicular skeletal muscle mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 52 | 109 | 48 | 47
gram | 447.96 (1688.08) | 538.45 (1224.13) | 464.75 (1513.96) | 632.18 (1928.68)

17. Secondary Outcome: Change in Lean Body Mass (Week 34)
Description: Change in Lean body mass was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 111 | 116
gram | 334.43 (2048.01) | 1359.33 (2359.11) | 1395.88 (2139.32)

18. Secondary Outcome: Change in Lean Body Mass (Week 87)
Description: Change in Lean body mass was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 52 | 109 | 48 | 47
gram | 1717.15 (2965.23) | 1719.87 (2515.90) | 1464.51 (2439.75) | 1681.82 (3413.61)

19. Secondary Outcome: Change in Bone Mineral Content (Week 87)
Description: Change in Bone mineral content was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 110 | 48 | 47
gram | -25.61 (93.35) | 5.02 (113.81) | -10.18 (99.18) | 32.33 (87.86)

20. Secondary Outcome: Change in Bone Mineral Density (Week 87)
Description: Change in Bone mineral density was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: grams per square centimeter
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 110 | 48 | 47
grams per square centimeter | -0.01 (0.04) | -0.00 (0.04) | -0.00 (0.04) | 0.01 (0.04)

21. Secondary Outcome: Change in IGF-I SDS (Week 34)
Description: Change in insulin-like growth factor (IGF-I) standard deviation scores (SDS) was measured from baseline (week -3) until the end of the main treatment period (week 34). A higher score reflects a better outcome.
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 113 | 116
Standard deviation score | 0.05 (0.59) | 2.28 (1.32) | 2.37 (1.33)

22. Secondary Outcome: Change in IGF-I SDS (Week 87)
Description: Change in IGF-I SDS was measured from baseline (week -3) until the end of the extension treatment period (week 87). A higher score reflects a better outcome.
Time Frame: Week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 47 | 47
Standard deviation score | 2.36 (1.55) | 2.29 (1.39) | 2.07 (1.12) | 2.35 (1.54)

23. Secondary Outcome: Change in IGFBP 3 SDS (Week 34)
Description: Change in insulin like growth factor binding protein 3 (IGFBP 3) SDS was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 113 | 116
Standard deviation score | 0.12 (0.61) | 1.44 (1.17) | 1.56 (1.24)

24. Secondary Outcome: Change in IGFBP 3 SDS (Week 87)
Description: Change in IGFBP 3 SDS was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: Week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 47 | 47
Standard deviation score | 1.33 (1.20) | 1.41 (1.20) | 1.30 (1.08) | 1.47 (1.51)

25. Secondary Outcome: Change in TRIM-AGHD (Total and Domain Scores) (Week 34)
Description: Change in treatment-related impact measure - adult growth hormone deficiency (TRIM-AGHD) scores (total and domain scores) was measured from baseline (week 0) until the end of the main treatment period (week 34). The TRIM-AGHD questionnaire measured the impact of GH treatment on the functioning and well-being of AGHD patients. The 4 concepts covered by the questionnaire were physical health, energy levels, cognitive ability and psychological health. TRIM-AGHD has 27 items and a total score as well as domain specific scores can be derived. The total score includes all answers that has been used to calculate each of the 4 subdomains. The score ranged from 0 to 100 for 'individual domains' and for the 'total', where a lower score reflected a better outcome.
Time Frame: Week 0, week 34
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Scores on a scale
  Energy: number analyzed (Participants) | 56 | 112 | 116
  Energy | -3.96 (25.40) | -13.42 (23.73) | -7.81 (24.07)
  Psychological: number analyzed (Participants) | 56 | 112 | 116
  Psychological | -3.38 (12.15) | -8.93 (14.21) | -4.63 (12.01)
  Cognitive: number analyzed (Participants) | 56 | 112 | 115
  Cognitive | -2.25 (18.17) | -7.06 (18.47) | -3.92 (17.29)
  Physical: number analyzed (Participants) | 56 | 112 | 115
  Physical | -5.88 (14.72) | -11.33 (19.23) | -7.39 (19.25)
  Total: number analyzed (Participants) | 56 | 112 | 115
  Total | -3.65 (12.05) | -9.99 (13.64) | -5.71 (12.69)

26. Secondary Outcome: Change in TRIM-AGHD (Total and Domain Scores) (Week 87)
Description: Change in TRIM-AGHD (total and domain scores) was measured from baseline (week 0) until the end of the extension treatment period (week 87). The TRIM-AGHD questionnaire measured the impact of GH treatment on the functioning and well-being of AGHD patients. The 4 concepts covered by the questionnaire were physical health, energy levels, cognitive ability and psychological health. TRIM-AGHD has 27 items and a total score as well as domain specific scores can be derived. The total score includes all answers that has been used to calculate each of the 4 subdomains. The score ranged from 0 to 100 for 'individual domains' and for the 'total', where a lower score reflected a better outcome.
Time Frame: week 0, week 87
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 61 | 120 | 52 | 51
Scores on scale
  Energy: number analyzed (Participants) | 54 | 111 | 49 | 47
  Energy | -11.73 (30.87) | -8.11 (25.46) | -23.30 (28.03) | -9.13 (26.98)
  Psychological: number analyzed (Participants) | 54 | 111 | 49 | 47
  Psychological | -6.97 (16.05) | -6.64 (14.56) | -15.64 (15.36) | -7.35 (10.50)
  Cognitive: number analyzed (Participants) | 54 | 111 | 49 | 48
  Cognitive | -4.88 (21.19) | -5.55 (18.59) | -14.18 (20.29) | -7.71 (14.14)
  Physical: number analyzed (Participants) | 54 | 111 | 49 | 48
  Physical | -11.19 (20.13) | -9.57 (21.94) | -17.22 (27.02) | -13.54 (18.02)
  Total: number analyzed (Participants) | 54 | 111 | 49 | 47
  Total | -8.28 (15.88) | -7.25 (14.42) | -17.38 (16.77) | -8.67 (11.73)

27. Secondary Outcome: Change in SF-36v2 (Summary and Domain Scores) (Week 34)
Description: SF-36v2™ questionnaire measured health-related quality of life (HRQoL) on 8 domains (Bodily Pain, General Health, Mental Health, Physical Functioning, Role Emotion, Physical Health, Social Functioning and Vitality) on individual scale ranges. The scores 0-100 (higher scores indicates better HRQoL) from SF-36 were converted to norm-based scores to enable a direct interpretation in relation to distribution of the scores in the 2009 U.S. general population. Mental component summary (MCS) measure is derived from domain scales of vitality, social functioning, role emotional and mental health. Physical component summary (PCS) measure is derived from domain scales of physical functioning, role-physical, bodily pain, and general health. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline.
Time Frame: Week 0, week 34
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Scores on scale
  Physical functioning: number analyzed (Participants) | 55 | 111 | 117
  Physical functioning | 2.19 (6.44) | 2.46 (7.08) | 3.18 (7.67)
  Role limitations due to physical health: number analyzed (Participants) | 56 | 111 | 117
  Role limitations due to physical health | 2.49 (7.68) | 3.95 (8.48) | 3.14 (9.06)
  Role limitations due to emotional health: number analyzed (Participants) | 56 | 111 | 117
  Role limitations due to emotional health | 2.29 (9.52) | 3.50 (10.87) | 3.06 (11.60)
  Vitality: number analyzed (Participants) | 56 | 111 | 118
  Vitality | 3.21 (7.67) | 5.26 (9.89) | 2.38 (8.56)
  Role limitations due to mental health: number analyzed (Participants) | 56 | 111 | 118
  Role limitations due to mental health | 0.85 (9.59) | 3.72 (10.17) | 2.78 (9.56)
  Social functioning: number analyzed (Participants) | 56 | 111 | 118
  Social functioning | 0.10 (10.43) | 3.19 (9.80) | 2.87 (9.69)
  Bodily pain: number analyzed (Participants) | 56 | 111 | 117
  Bodily pain | 0.63 (8.79) | 2.19 (9.50) | 1.79 (9.52)
  General health: number analyzed (Participants) | 56 | 111 | 118
  General health | 1.50 (7.25) | 4.47 (7.64) | 1.85 (7.58)
  Overall physical: number analyzed (Participants) | 55 | 111 | 116
  Overall physical | 2.01 (6.22) | 2.87 (6.33) | 2.40 (6.53)
  Overall mental: number analyzed (Participants) | 55 | 111 | 116
  Overall mental | 1.28 (8.72) | 4.09 (10.19) | 2.70 (9.29)

28. Secondary Outcome: Change in SF-36v2 (Summary and Domain Scores) (Week 87)
Description: as for outcome 27
Time Frame: week 0, week 87
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 61 | 120 | 52 | 51
Score on scale
  Physical functioning: number analyzed (Participants) | 53 | 111 | 49 | 48
  Physical functioning | 2.87 (8.13) | 3.83 (7.66) | 3.43 (6.96) | 1.84 (8.07)
  Role limitations due to physical health: number analyzed (Participants) | 54 | 110 | 49 | 48
  Role limitations due to physical health | 3.31 (9.81) | 4.16 (10.10) | 4.65 (10.06) | 2.45 (10.50)
  Role limitations due to emotional health: number analyzed (Participants) | 54 | 110 | 49 | 48
  Role limitations due to emotional health | 3.46 (11.59) | 3.46 (12.25) | 7.30 (13.46) | 1.13 (11.20)
  Vitality: number analyzed (Participants) | 54 | 111 | 49 | 48
  Vitality | 6.71 (11.01) | 4.18 (9.30) | 8.16 (12.77) | 4.16 (8.88)
  Role limitations due to mental health: number analyzed (Participants) | 54 | 111 | 49 | 48
  Role limitations due to mental health | 2.80 (10.55) | 3.66 (8.12) | 6.12 (13.02) | 1.70 (10.31)
  Social functioning: number analyzed (Participants) | 54 | 111 | 49 | 48
  Social functioning | 3.84 (10.36) | 3.44 (10.29) | 4.56 (10.34) | 0.57 (11.26)
  Bodily pain: number analyzed (Participants) | 54 | 110 | 49 | 48
  Bodily pain | 1.41 (8.57) | 1.47 (10.29) | 3.51 (9.57) | 0.30 (11.25)
  General health: number analyzed (Participants) | 54 | 111 | 49 | 48
  General health | 3.46 (7.33) | 3.32 (7.70) | 5.66 (9.67) | 2.20 (8.66)
  Overall physical score: number analyzed (Participants) | 53 | 109 | 49 | 48
  Overall physical score | 2.66 (6.91) | 2.98 (7.24) | 3.06 (7.07) | 1.81 (7.72)
  Overall mental score: number analyzed (Participants) | 53 | 109 | 49 | 48
  Overall mental score | 4.51 (10.39) | 3.56 (9.06) | 7.50 (13.59) | 1.66 (10.18)

29. Secondary Outcome: TSQM-9 Scores (Domain Scores) (Week 34)
Description: Scores from the TSQM-9 scale were calculated at the end of the main treatment period (week 34). The Treatment Satisfaction Questionnaire for Medication - 9 items (TSQM-9) is a generic questionnaire that measures a patients' satisfaction with medication. Items are rated on a 5-point or 7-point scale according to patients' experience with the medication. The items covered are satisfaction with the effect of the medication, convenience and global treatment satisfaction. Each domain is based on 3 questions. The score is calculated in a range from 0 to 100, where a higher score reflects a better outcome. Scores have been summed and then scaled to 0-100.
Time Frame: Week 34
Population: Overall number of participants analyzed = FAS. Number analyzed = Number of participants with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Scores on a scale
  Effectiveness: number analyzed (Participants) | 55 | 110 | 118
  Effectiveness | 49.6 (22.2) | 67.1 (21.8) | 56.1 (22.5)
  Convenience: number analyzed (Participants) | 55 | 111 | 118
  Convenience | 74.3 (16.9) | 73.9 (18.7) | 77.7 (15.3)
  Global satisfaction: number analyzed (Participants) | 55 | 110 | 118
  Global satisfaction | 54.0 (24.8) | 69.0 (24.0) | 63.1 (24.2)

30. Secondary Outcome: TSQM-9 Scores (Domain Scores) (Week 87)
Description: Scores from the TSQM-9 scale were calculated at the end of the extension treatment period (week 87). The Treatment Satisfaction Questionnaire for Medication - 9 items (TSQM-9) is a generic questionnaire that measures a patients' satisfaction with medication. Items are rated on a 5-point or 7-point scale according to patients' experience with the medication. The items covered are satisfaction with the effect of the medication, convenience and global treatment satisfaction. Each domain is based on 3 questions. The score is calculated in a range from 0 to 100, where a higher score reflects a better outcome. Scores have been summed and then scaled to 0-100.
Time Frame: Week 87
Population: Overall number of participants analyzed = FAS. Number analyzed = Number of participants with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 61 | 120 | 52 | 51
Scores on a scale
  Effectiveness: number analyzed (Participants) | 54 | 111 | 49 | 49
  Effectiveness | 59.7 (23.1) | 65.7 (22.4) | 69.6 (24.0) | 70.9 (20.9)
  Convenience: number analyzed (Participants) | 61 | 120 | 52 | 49
  Convenience | 75.1 (19.1) | 80.0 (16.5) | 72.6 (20.0) | 79.4 (17.1)
  Global satisfaction: number analyzed (Participants) | 61 | 120 | 52 | 49
  Global satisfaction | 63.2 (26.2) | 68.1 (24.6) | 71.7 (25.3) | 75.1 (23.6)

31. Secondary Outcome: Change in Total Cholesterol (Week 34)
Description: Change in Total cholesterol was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 119
mmol/L | 0.03 (0.96) | -0.10 (0.91) | -0.09 (0.78)

32. Secondary Outcome: Change in Total Cholesterol (Week 87)
Description: Change in Total cholesterol was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | -0.21 (0.89) | 0.03 (0.96) | -0.05 (0.94) | -0.33 (1.08)

33. Secondary Outcome: Change in HDL-cholesterol (Week 34)
Description: Change in High-density lipoprotein (HDL) cholesterol was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 119
mmol/L | -0.00 (0.37) | 0.02 (0.28) | 0.05 (0.30)

34. Secondary Outcome: Change in HDL-cholesterol (Week 87)
Description: Change in HDL-cholesterol was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | 0.06 (0.30) | 0.05 (0.32) | 0.09 (0.27) | 0.06 (0.34)

35. Secondary Outcome: Change in LDL-cholesterol (Week 34)
Description: Change in Low-density lipoprotein (LDL) cholesterol was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 119
mmol/L | 0.02 (0.75) | -0.18 (0.72) | -0.13 (0.64)

36. Secondary Outcome: Change in LDL-cholesterol (Week 87)
Description: Change in LDL-cholesterol was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | -0.30 (0.72) | -0.06 (0.81) | -0.15 (0.85) | -0.36 (0.90)

37. Secondary Outcome: Change in Triglycerides (Week 34)
Description: Change in Triglycerides was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 119
mmol/L | 0.01 (0.65) | 0.13 (0.62) | -0.02 (0.73)

38. Secondary Outcome: Change in Triglycerides (Week 87)
Description: Change in Triglycerides was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | 0.07 (0.48) | 0.03 (0.76) | 0.03 (0.56) | -0.08 (0.73)

39. Secondary Outcome: Change in Hs-CRP (Week 34)
Description: Change in high-sensitivity C-reactive protein (hs-CRP) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 116
mg/L | 0.405 (13.144) | -1.604 (13.254) | -0.569 (5.616)

40. Secondary Outcome: Change in Hs-CRP (Week 87)
Description: Change in hs-CRP was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 111 | 49 | 49
mg/L | -0.325 (16.247) | -1.445 (3.791) | -0.857 (17.491) | -1.257 (12.497)

41. Secondary Outcome: Change in IL-6 (Week 34)
Description: Change in Interleukin 6 (IL-6) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 113 | 118
pg/mL | 3.48 (24.84) | 0.07 (4.01) | 0.18 (5.78)

42. Secondary Outcome: Change in IL-6 (Week 87)
Description: Change in IL-6 was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 111 | 48 | 47
pg/mL | 0.11 (3.30) | 0.52 (6.19) | 0.49 (5.12) | 1.19 (2.92)

43. Secondary Outcome: Change in Body Weight (Week 34)
Description: Change in body weight was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 119
Kg | 0.6 (2.9) | 0.2 (4.0) | 1.3 (4.2)

44. Secondary Outcome: Change in Body Weight (Week 87)
Description: Change in body weight was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
Kg | 1.2 (4.4) | 1.4 (4.8) | 0.4 (5.2) | 2.1 (7.0)

45. Secondary Outcome: Change in Waist Circumference (Week 34)
Description: Change in waist circumference was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 55 | 113 | 117
cm | 0.82 (4.50) | -0.66 (4.83) | -0.00 (4.52)

46. Secondary Outcome: Change in Waist Circumference (Week 87)
Description: Change in waist circumference was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 111 | 49 | 49
cm | 1.35 (5.62) | 0.53 (5.17) | -2.26 (7.93) | 0.74 (7.17)

47. Secondary Outcome: Number of Adverse Events (Weeks 0-35)
Description: Number of adverse events from baseline (week 0) until the end of week 35 were reported. This endpoint shows number of treatment-emergent adverse events (TEAEs), including the injection site reactions.
Time Frame: Weeks 0-35
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Events | 184 | 426 | 385

48. Secondary Outcome: Number of Adverse Events (Weeks 0-88)
Description: Number of adverse events from baseline (week 0) until the end of week 88 were reported. This endpoint shows the number of TEAEs along with the injection site reactions.
Time Frame: Weeks 0-88
Population: as for outcome 47
Measure: Number; unit: Events
Groups:
- Norditropin/-: Participants who received Norditropin in the main period of the trial and discontinued after the main period of the study are included here.
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan | Norditropin/-
Number analyzed (Participants) | 61 | 120 | 52 | 51 | 16
Events | 395 | 699 | 384 | 385 | 49

49. Secondary Outcome: Occurrence of Anti-NNC0195-0092 Antibodies (Weeks 0-35)
Description: Number of participants with anti-NNC0195-0092 antibodies at week 35 was recorded. The numbers presented in this endpoint are the participants that were found to have positive antibodies.
Time Frame: Weeks 0 to 35
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 109 | 120
Participants | 0 | 1 | 0

50. Secondary Outcome: Occurrence of Anti-NNC0195-0092 Antibodies (Weeks 0-88)
Description: Number of participants with anti-NNC0195-0092 antibodies at week 88 was recorded. The numbers presented in this endpoint are the participants that were found to have positive antibodies.
Time Frame: Weeks 0 to 88
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan | Norditropin/-
Number analyzed (Participants) | 61 | 120 | 52 | 51 | 16
Participants | 0 | 0 | 0 | 0 | 1

51. Secondary Outcome: Incidence of Technical Complaints During Exposure to Trial Product (Weeks 0-35)
Description: Incidence of technical complaints were recorded from baseline (week 0) until week 35.
Time Frame: Weeks 0 to 35
Population: as for outcome 47
Measure: Number; unit: Technical complaints
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Technical complaints | 1 | 14 | 0

52. Secondary Outcome: Incidence of Technical Complaints During Exposure to Trial Product (Weeks 0-88)
Description: Incidence of technical complaints were recorded from baseline (week 0) until week 88.
Time Frame: Weeks 0 to 88
Population: as for outcome 47
Measure: Number; unit: Technical complaints
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 61 | 120 | 52 | 51
Technical complaints | 1 | 6 | 18 | 7

53. Secondary Outcome: Change in Physical Examination During Exposure to Trial Product (Week 35)
Description: Change in physical examination from baseline (week 0) until the end of the main treatment period (week 35) was reported. Results are presented for the following examinations: 1) Head, neck, eyes and nose 2) Respiratory system (sys.) 3) Cardiovascular sys. 4) Gastrointestinal sys. 5) Musculoskeletal sys. 6) Central & Peripheral nervous sys. 7) Skin 8) Lymph node palpation
Time Frame: Week 0 and week 35
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Participants
  Head, neck, eyes, nose (Week 0): Normal | 55 | 111 | 108
  Head, neck, eyes, nose (Week 0): Abnormal, not clinically significant (NCS) | 6 | 6 | 7
  Head, neck, eyes, nose (Week 0): Abnormal, clinically significant (CS) | 0 | 2 | 5
  Head, neck, eyes, nose (Week 0): Missing | 0 | 0 | 0
  Head, neck, eyes, nose (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Head, neck, eyes, nose (Week 35): Normal | 51 | 98 | 107
  Head, neck, eyes, nose (Week 35): Abnormal, not clinically significant (NCS) | 5 | 4 | 9
  Head, neck, eyes, nose (Week 35): Abnormal, clinically significant (CS) | 0 | 3 | 2
  Head, neck, eyes, nose (Week 35): Missing | 0 | 0 | 0
  Respiratory sys. (Week 0): Normal | 61 | 118 | 119
  Respiratory sys. (Week 0): Abnormal, not clinically significant (NCS) | 0 | 1 | 1
  Respiratory sys. (Week 0): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Respiratory sys. (Week 0): Missing | 0 | 0 | 0
  Respiratory sys. (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Respiratory sys. (Week 35): Normal | 56 | 103 | 117
  Respiratory sys. (Week 35): Abnormal, not clinically significant (NCS) | 0 | 2 | 1
  Respiratory sys. (Week 35): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Respiratory sys. (Week 35): Missing | 0 | 0 | 0
  Cardiovascular sys. (Week 0): Normal | 56 | 112 | 116
  Cardiovascular sys. (Week 0): Abnormal, not clinically significant (NCS) | 4 | 7 | 4
  Cardiovascular sys. (Week 0): Abnormal, clinically significant (CS) | 1 | 0 | 0
  Cardiovascular sys. (Week 0): Missing | 0 | 0 | 0
  Cardiovascular sys. (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Cardiovascular sys. (Week 35): Normal | 54 | 99 | 112
  Cardiovascular sys. (Week 35): Abnormal, not clinically significant (NCS) | 1 | 6 | 6
  Cardiovascular sys. (Week 35): Abnormal, clinically significant (CS) | 1 | 0 | 0
  Cardiovascular sys. (Week 35): Missing | 0 | 0 | 0
  Gastrointestinal sys. (Week 0): Normal | 59 | 113 | 119
  Gastrointestinal sys. (Week 0): Abnormal, not clinically significant (NCS) | 2 | 6 | 1
  Gastrointestinal sys. (Week 0): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Gastrointestinal sys. (Week 0): Missing | 0 | 0 | 0
  Gastrointestinal sys. (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Gastrointestinal sys. (Week 35): Normal | 53 | 98 | 116
  Gastrointestinal sys. (Week 35): Abnormal, not clinically significant (NCS) | 3 | 7 | 2
  Gastrointestinal sys. (Week 35): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Gastrointestinal sys. (Week 35): Missing | 0 | 0 | 0
  Musculoskeletal sys. (Week 0): Normal | 59 | 111 | 113
  Musculoskeletal sys. (Week 0): Abnormal, not clinically significant (NCS) | 2 | 6 | 5
  Musculoskeletal sys. (Week 0): Abnormal, clinically significant (CS) | 0 | 2 | 2
  Musculoskeletal sys. (Week 0): Missing | 0 | 0 | 0
  Musculoskeletal sys. (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Musculoskeletal sys. (Week 35): Normal | 54 | 96 | 111
  Musculoskeletal sys. (Week 35): Abnormal, not clinically significant (NCS) | 2 | 7 | 5
  Musculoskeletal sys. (Week 35): Abnormal, clinically significant (CS) | 0 | 2 | 2
  Musculoskeletal sys. (Week 35): Missing | 0 | 0 | 0
  Central & Peripheral nervous sys (Week 0): Normal | 59 | 113 | 117
  Central & Peripheral nervous sys (Week 0): Abnormal, not clinically significant (NCS) | 2 | 5 | 3
  Central & Peripheral nervous sys (Week 0): Abnormal, clinically significant (CS) | 0 | 1 | 0
  Central & Peripheral nervous sys (Week 0): Missing | 0 | 0 | 0
  Central & Peripheral nervous sys (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Central & Peripheral nervous sys (Week 35): Normal | 55 | 101 | 114
  Central & Peripheral nervous sys (Week 35): Abnormal, not clinically significant (NCS) | 1 | 4 | 4
  Central & Peripheral nervous sys (Week 35): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Central & Peripheral nervous sys (Week 35): Missing | 0 | 0 | 0
  Skin (Week 0): Normal | 51 | 100 | 109
  Skin (Week 0): Abnormal, not clinically significant (NCS) | 9 | 17 | 11
  Skin (Week 0): Abnormal, clinically significant (CS) | 1 | 2 | 0
  Skin (Week 0): Missing | 0 | 0 | 0
  Skin (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Skin (Week 35): Normal | 51 | 88 | 102
  Skin (Week 35): Abnormal, not clinically significant (NCS) | 5 | 15 | 13
  Skin (Week 35): Abnormal, clinically significant (CS) | 0 | 2 | 3
  Skin (Week 35): Missing | 0 | 0 | 0
  Lymph node palpation (Week 0): Normal | 61 | 119 | 120
  Lymph node palpation (Week 0): Abnormal, not clinically significant (NCS) | 0 | 0 | 0
  Lymph node palpation (Week 0): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Lymph node palpation (Week 0): Missing | 0 | 0 | 0
  Lymph node palpation (Week 35): number analyzed (Participants) | 56 | 105 | 118
  Lymph node palpation (Week 35): Normal | 56 | 105 | 118
  Lymph node palpation (Week 35): Abnormal, not clinically significant (NCS) | 0 | 0 | 0
  Lymph node palpation (Week 35): Abnormal, clinically significant (CS) | 0 | 0 | 0
  Lymph node palpation (Week 35): Missing | 0 | 0 | 0

54. Secondary Outcome: Change in Physical Examination During Exposure to Trial Product (Week 88)
Description: Change in physical examination from baseline (week 0) until the end of the extension period (week 88) was reported. Results are presented for the following examinations: 1) Head, neck, eyes and nose 2) Respiratory system (sys.) 3) Cardiovascular sys. 4) Gastrointestinal sys. 5) Musculoskeletal sys. 6) Central & Peripheral nervous sys. 7) Skin 8) Lymph node palpation
Time Frame: Week 0 and week 88
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan | Norditropin/-
Number analyzed (Participants) | 61 | 120 | 52 | 51 | 16
Participants
  Head, neck, eyes, nose (Week 0): Normal | 55 | 108 | 49 | 47 | 15
  Head, neck, eyes, nose (Week 0): Abnormal, NCS | 6 | 7 | 2 | 3 | 1
  Head, neck, eyes, nose (Week 0): Abnormal, CS | 0 | 5 | 1 | 1 | 0
  Head, neck, eyes, nose (Week 0): Missing | 0 | 0 | 0 | 0 | 0
  Head, neck, eyes, nose (Week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Head, neck, eyes, nose (Week 88): Normal | 48 | 101 | 46 | 44 | 0
  Head, neck, eyes, nose (Week 88): Abnormal, NCS | 6 | 7 | 2 | 1 | 0
  Head, neck, eyes, nose (Week 88): Abnormal, CS | 0 | 1 | 1 | 3 | 0
  Head, neck, eyes, nose (Week 88): Missing | 0 | 1 | 0 | 0 | 0
  Respiratory sys. (Week 0): Normal | 61 | 119 | 52 | 50 | 16
  Respiratory sys. (Week 0): Abnormal, NCS | 0 | 1 | 0 | 1 | 0
  Respiratory sys. (Week 0): Abnormal, CS | 0 | 0 | 0 | 0 | 0
  Respiratory sys. (Week 0): Missing | 0 | 0 | 0 | 0 | 0
  Respiratory sys. (Week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Respiratory sys. (Week 88): Normal | 54 | 109 | 49 | 47 | 0
  Respiratory sys. (Week 88): Abnormal, NCS | 0 | 0 | 0 | 1 | 0
  Respiratory sys. (Week 88): Abnormal, CS | 0 | 0 | 0 | 0 | 0
  Respiratory sys. (Week 88): Missing | 0 | 1 | 0 | 0 | 0
  Cardiovascular sys. (Week 0): Normal | 56 | 116 | 49 | 47 | 16
  Cardiovascular sys. (Week 0): Abnormal, NCS | 4 | 4 | 3 | 4 | 0
  Cardiovascular sys. (Week 0): Abnormal, CS | 1 | 0 | 0 | 0 | 0
  Cardiovascular sys. (Week 0): Missing | 0 | 0 | 0 | 0 | 0
  Cardiovascular sys. (Week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Cardiovascular sys. (Week 88): Normal | 52 | 107 | 45 | 47 | 0
  Cardiovascular sys. (Week 88): Abnormal, NCS | 1 | 2 | 4 | 1 | 0
  Cardiovascular sys. (Week 88): Abnormal, CS | 1 | 0 | 0 | 0 | 0
  Cardiovascular sys. (Week 88): Missing | 0 | 1 | 0 | 0 | 0
  Gastrointestinal sys. (Week 0): Normal | 59 | 119 | 49 | 49 | 15
  Gastrointestinal sys. (Week 0): Abnormal, NCS | 2 | 1 | 3 | 2 | 1
  Gastrointestinal sys. (Week 0): Abnormal, CS | 0 | 0 | 0 | 0 | 0
  Gastrointestinal sys. (Week 0): Missing | 0 | 0 | 0 | 0 | 0
  Gastrointestinal sys. (Week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Gastrointestinal sys. (Week 88): Normal | 52 | 109 | 47 | 48 | 0
  Gastrointestinal sys. (Week 88): Abnormal, NCS | 2 | 0 | 2 | 0 | 0
  Gastrointestinal sys. (Week 88): Abnormal, CS | 0 | 0 | 0 | 0 | 0
  Gastrointestinal sys. (Week 88): Missing | 0 | 1 | 0 | 0 | 0
  Musculoskeletal sys. (Week 0): Normal | 59 | 113 | 48 | 49 | 14
  Musculoskeletal sys. (Week 0): Abnormal, NCS | 2 | 5 | 2 | 2 | 2
  Musculoskeletal sys. (Week 0): Abnormal, CS | 0 | 2 | 2 | 0 | 0
  Musculoskeletal sys. (Week 0): Missing | 0 | 0 | 0 | 0 | 0
  Musculoskeletal sys. (Week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Musculoskeletal sys. (Week 88): Normal | 49 | 101 | 45 | 46 | 0
  Musculoskeletal sys. (Week 88): Abnormal, NCS | 4 | 7 | 3 | 2 | 0
  Musculoskeletal sys. (Week 88): Abnormal, CS | 1 | 1 | 1 | 0 | 0
  Musculoskeletal sys. (Week 88): Missing | 0 | 1 | 0 | 0 | 0
  Central & Peripheral nervous sys. (week 0): Normal | 59 | 117 | 51 | 48 | 14
  Central & Peripheral nervous sys. (week 0): Abnormal, NCS | 2 | 3 | 1 | 3 | 1
  Central & Peripheral nervous sys. (week 0): Abnormal, CS | 0 | 0 | 0 | 0 | 1
  Central & Peripheral nervous sys. (week 0): Missing | 0 | 0 | 0 | 0 | 0
  Central & Peripheral nervous sys. (week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Central & Peripheral nervous sys. (week 88): Normal | 53 | 106 | 49 | 45 | 0
  Central & Peripheral nervous sys. (week 88): Abnormal, NCS | 1 | 3 | 0 | 3 | 0
  Central & Peripheral nervous sys. (week 88): Abnormal, CS | 0 | 0 | 0 | 0 | 0
  Central & Peripheral nervous sys. (week 88): Missing | 0 | 1 | 0 | 0 | 0
  Skin (Week 0): Normal | 51 | 109 | 48 | 41 | 11
  Skin (Week 0): Abnormal, NCS | 9 | 11 | 3 | 10 | 4
  Skin (Week 0): Abnormal, CS | 1 | 0 | 1 | 0 | 1
  Skin (Week 0): Missing | 0 | 0 | 0 | 0 | 0
  Skin (Week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Skin (Week 88): Normal | 49 | 96 | 42 | 42 | 0
  Skin (Week 88): Abnormal, NCS | 3 | 8 | 6 | 5 | 0
  Skin (Week 88): Abnormal, CS | 2 | 5 | 1 | 1 | 0
  Skin (Week 88): Missing | 0 | 1 | 0 | 0 | 0
  Lymph node palpation (week 0): Normal | 61 | 120 | 52 | 51 | 16
  Lymph node palpation (week 0): Abnormal, NCS | 0 | 0 | 0 | 0 | 0
  Lymph node palpation (week 0): Abnormal, CS | 0 | 0 | 0 | 0 | 0
  Lymph node palpation (week 0): Missing | 0 | 0 | 0 | 0 | 0
  Lymph node palpation (week 88): number analyzed (Participants) | 54 | 110 | 49 | 48 | 0
  Lymph node palpation (week 88): Normal | 53 | 108 | 49 | 48 | 0
  Lymph node palpation (week 88): Abnormal, NCS | 0 | 1 | 0 | 0 | 0
  Lymph node palpation (week 88): Abnormal, CS | 1 | 0 | 0 | 0 | 0
  Lymph node palpation (week 88): Missing | 0 | 1 | 0 | 0 | 0

55. Secondary Outcome: Change in Electrocardiogram (ECG) Evaluation During Exposure to Trial Product (Week 35)
Description: Change in Electrocardiogram (ECG) evaluation from baseline (week -3) until the end of the main treatment period (week 35) was reported.
Time Frame: Week -3 and week 35
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 61 | 119 | 120
Participants
  Week -3: Normal | 30 | 67 | 77
  Week -3: Abnormal, NCS | 29 | 52 | 40
  Week -3: Abnormal, CS | 2 | 0 | 3
  Week -3: Missing | 0 | 0 | 0
  Week 35: number analyzed (Participants) | 57 | 111 | 119
  Week 35: Normal | 29 | 65 | 77
  Week 35: Abnormal, NCS | 26 | 42 | 34
  Week 35: Abnormal, CS | 1 | 0 | 2
  Week 35: Missing | 1 | 4 | 6

56. Secondary Outcome: Change in ECG Evaluation During Exposure to Trial Product (Week 88)
Description: Change in ECG evaluation from baseline (week 0) until the end of the extension period (Week 88) was reported.
Time Frame: Week -3 and week 88
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan | Norditropin/-
Number analyzed (Participants) | 61 | 120 | 52 | 51 | 16
Participants
  Week -3: Normal | 30 | 77 | 26 | 34 | 7
  Week -3: Abnormal, NCS | 29 | 40 | 26 | 17 | 9
  Week -3: Abnormal, CS | 2 | 3 | 0 | 0 | 0
  Week -3: Missing | 0 | 0 | 0 | 0 | 0
  Week 88: number analyzed (Participants) | 54 | 109 | 49 | 49 | 1
  Week 88: Normal | 34 | 74 | 29 | 35 | 0
  Week 88: Abnormal, NCS | 18 | 34 | 18 | 12 | 0
  Week 88: Abnormal, CS | 1 | 1 | 2 | 1 | 0
  Week 88: Missing | 1 | 0 | 0 | 1 | 1

57. Secondary Outcome: Change in Diastolic Blood Pressure (Week 35)
Description: Change in diastolic blood pressure was measured from baseline (week -3) until the end of the main treatment period (week 35).
Time Frame: Week -3, week 35
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 107 | 118
mm Hg | -0.41 (7.75) | -2.07 (8.73) | -1.42 (8.98)

58. Secondary Outcome: Change in Diastolic Blood Pressure (Week 88)
Description: Change in diastolic blood pressure was measured from baseline (week -3) until the end of the extension treatment period week 88.
Time Frame: Week -3, week 88
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 49 | 48
mm Hg | -2.48 (7.77) | -0.85 (9.21) | -0.61 (8.71) | -2.10 (9.50)

59. Secondary Outcome: Change in Systolic Blood Pressure (Week 35)
Description: Change in systolic blood pressure was measured from baseline (week -3) until the end of the main treatment period (week 35).
Time Frame: Week -3, week 35
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 107 | 118
mm Hg | 1.13 (11.35) | -2.81 (13.33) | -1.39 (12.89)

60. Secondary Outcome: Change in Systolic Blood Pressure (Week 88)
Description: Change in systolic blood pressure was measured from baseline (week -3) until the end of the extension treatment period (week 88).
Time Frame: Week -3, week 88
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 49 | 48
mm Hg | -1.30 (12.18) | 0.45 (13.01) | -1.35 (13.07) | -1.83 (11.63)

61. Secondary Outcome: Change in Pulse (Week 35)
Description: Change in pulse was measured from baseline (week -3) until the end of the main treatment period (week 35).
Time Frame: Week -3, week 35
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 119
beats/min | 0.54 (9.43) | 2.61 (9.74) | 1.02 (10.20)

62. Secondary Outcome: Change in Pulse (Week 88)
Description: Change in pulse was measured from baseline (week -3) until the end of the extension treatment period (week 88).
Time Frame: Week -3, week 88
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 49 | 48
beats/min | 0.78 (11.70) | -0.55 (10.51) | -0.55 (10.32) | 0.08 (8.75)

63. Secondary Outcome: Change in Haemoglobin (Week 34)
Description: Change in Haemoglobin was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 119
g/L | 1.87 (10.25) | -0.51 (8.80) | 0.64 (8.78)

64. Secondary Outcome: Change in Haemoglobin (Week 87)
Description: Change in Haemoglobin was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 109 | 48 | 48
g/L | 2.93 (11.36) | 2.76 (9.54) | -0.40 (9.22) | 0.86 (15.96)

65. Secondary Outcome: Change in Haematocrit (Week 34)
Description: Change in Haematocrit was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: % of red blood cells
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 119
% of red blood cells | 0.5 (3.3) | -0.3 (2.9) | 0.1 (3.1)

66. Secondary Outcome: Change in Haematocrit (Week 87)
Description: Change in Haematocrit was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: % of red blood cells
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 109 | 48 | 48
% of red blood cells | 0.17 (3.44) | 0.21 (3.29) | -0.59 (2.78) | -0.48 (5.10)

67. Secondary Outcome: Change in Erythrocytes (Week 34)
Description: Change in Erythrocytes was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cells/pL
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 119
cells/pL | 0.09 (0.33) | 0.06 (0.29) | 0.08 (0.32)

68. Secondary Outcome: Change in Erythrocytes (Week 87)
Description: Change in Erythrocytes was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cells/pL
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 109 | 48 | 48
cells/pL | 0.09 (0.34) | 0.12 (0.35) | 0.01 (0.31) | 0.05 (0.54)

69. Secondary Outcome: Change in Mean Corpuscular Volume (MCV) (Week 34)
Description: Change in Mean corpuscular volume (MCV) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 119
fL | -0.6 (3.3) | -1.8 (3.6) | -1.5 (3.0)

70. Secondary Outcome: Change in Mean Corpuscular Volume (MCV) (Week 87)
Description: Change in Mean corpuscular volume (MCV) was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 109 | 48 | 48
fL | -1.39 (4.27) | -1.80 (3.31) | -1.31 (3.63) | -1.77 (3.66)

71. Secondary Outcome: Change in Mean Corpuscular Haemoglobin Concentration (MCHC) (Week 34)
Description: Change in Mean corpuscular haemoglobin concentration (MCHC) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 119
mmol/L | 0.1 (0.5) | 0.1 (0.6) | 0.1 (0.6)

72. Secondary Outcome: Change in Mean Corpuscular Haemoglobin Concentration (MCHC) (Week 87)
Description: Change in Mean corpuscular haemoglobin concentration (MCHC) was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 109 | 48 | 48
mmol/L | 0.36 (0.47) | 0.29 (0.61) | 0.23 (0.70) | 0.35 (0.52)

73. Secondary Outcome: Change in Thrombocytes (Week 34)
Description: Change in Thrombocytes was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 111 | 115
10^9 cells/L | 1.6 (37.4) | 10.8 (37.1) | 15.3 (35.0)

74. Secondary Outcome: Change in Thrombocytes (Week 87)
Description: Change in Thrombocytes was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 108 | 47 | 48
10^9 cells/L | -1.2 (44.7) | 11.0 (36.7) | -0.9 (31.3) | 6.6 (53.4)

75. Secondary Outcome: Change in Leucocytes (Week 34)
Description: Change in Leucocytes was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 119
10^9 cells/L | 0.22 (1.57) | -0.05 (1.50) | -0.32 (1.75)

76. Secondary Outcome: Change in Leucocytes (Week 87)
Description: Change in Leucocytes was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 109 | 48 | 48
10^9 cells/L | 0.29 (1.93) | -0.12 (1.94) | -0.14 (1.44) | -0.14 (2.55)

77. Secondary Outcome: Change in Alanine Aminotransferase (ALT) (Week 34)
Description: Change in ALT was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
U/L | 4.5 (24.7) | -1.4 (11.9) | -4.4 (17.9)

78. Secondary Outcome: Change in Alanine Aminotransferase (ALT) (Week 87)
Description: Change in ALT was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
U/L | -1.1 (13.1) | -4.3 (16.9) | 0.6 (12.5) | -3.0 (14.6)

79. Secondary Outcome: Change in Albumin (Week 34)
Description: Change in Albumin was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
g/L | 6.09 (3.56) | -0.72 (2.81) | -0.42 (3.06)

80. Secondary Outcome: Change in Albumin (Week 87)
Description: Change in Albumin was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
g/L | -1.19 (3.15) | -0.86 (3.12) | -1.12 (3.52) | -1.69 (3.01)

81. Secondary Outcome: Change in Alkaline Phosphatase (ALP) (Week 34)
Description: Change in Alkaline phosphatase (ALP) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 118
U/L | 1.8 (16.5) | 7.9 (24.3) | 5.8 (14.9)

82. Secondary Outcome: Change in Alkaline Phosphatase (AP) (Week 87)
Description: Change in Alkaline phosphatase (AP) was measured from baseline (week -3) until the end of the week 87.
Time Frame: Week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 48 | 49
U/L | 8.1 (20.2) | 5.4 (16.0) | 3.3 (22.2) | 4.2 (18.0)

83. Secondary Outcome: Change in Aspartate Aminotransferase (AST) (Week 34)
Description: Change in AST was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
U/L | 1.96 (15.11) | -0.80 (9.38) | -2.00 (13.97)

84. Secondary Outcome: Change in Aspartate Aminotransferase (AST) (Week 87)
Description: Change in AST was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: Week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
U/L | 1.76 (24.346) | -2.17 (13.98) | -0.43 (5.94) | -1.69 (12.75)

85. Secondary Outcome: Change in Bilirubin (Week 34)
Description: Change in Bilirubin was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
umol/L | -0.08 (4.76) | -0.38 (4.10) | -0.41 (4.09)

86. Secondary Outcome: Change in Bilirubin (Week 87)
Description: Change in Bilirubin was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 111 | 47 | 48
umol/L | 0.04 (3.77) | 0.14 (4.45) | 0.45 (3.24) | -0.33 (4.52)

87. Secondary Outcome: Change in Calcium (Week 34)
Description: Change in Calcium was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 112 | 118
mmol/L | 0.00 (0.13) | 0.04 (0.14) | 0.03 (0.11)

88. Secondary Outcome: Change in Calcium (Week 87)
Description: Change in Calcium was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | 0.01 (0.12) | 0.03 (0.12) | 0.03 (0.11) | 0.01 (0.12)

89. Secondary Outcome: Change in Chloride (Week 34)
Description: Change in Chloride was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
mmol/L | -1.1 (2.7) | -0.6 (2.9) | -0.3 (2.9)

90. Secondary Outcome: Change in Chloride (Week 87)
Description: Change in Chloride was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | -1.8 (3.5) | -1.0 (3.0) | -1.1 (3.2) | -0.6 (3.1)

91. Secondary Outcome: Change in Creatinine (Week 34)
Description: Change in Creatinine was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
umol/L | 0.9 (9.4) | -2.8 (10.9) | -2.9 (10.6)

92. Secondary Outcome: Change in Creatinine (Week 87)
Description: Change in Creatinine was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
umol/L | -5.6 (11.9) | -2.5 (11.7) | -2.0 (9.8) | 1.8 (41.2)

93. Secondary Outcome: Change in Creatine Kinase (Week 34)
Description: Change in Creatine kinase was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
U/L | 5.0 (136.6) | 10.9 (101.0) | -23.5 (355.0)

94. Secondary Outcome: Change in Creatine Kinase (Week 87)
Description: Change in Creatine kinase was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
U/L | 228.7 (1603.3) | -9.4 (411.3) | 1.3 (89.3) | 30.5 (125.7)

95. Secondary Outcome: Change in Gamma-glutamyl Transferase (GGT) (Week 34)
Description: Change in GGT was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
U/L | 9.3 (66.2) | -5.8 (17.0) | -4.2 (27.5)

96. Secondary Outcome: Change in Gamma-glutamyl Transferase (GGT) (Week 87)
Description: Change in GGT was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
U/L | 19.4 (16.4) | 29.3 (39.3) | 25.9 (23.8) | 20.7 (13.9)

97. Secondary Outcome: Change in Phosphate (Inorganic) (Week 34)
Description: Change in Phosphate (inorganic) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
mmol/L | -0.038 (0.183) | 0.155 (0.182) | 0.181 (0.202)

98. Secondary Outcome: Change in Phosphate (Inorganic)(Week 87)
Description: Change in Phosphate (inorganic) was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | 0.100 (0.190) | 0.125 (0.193) | 0.076 (0.190) | 0.115 (0.219)

99. Secondary Outcome: Change in Potassium (Week 34)
Description: Change in Potassium was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 52 | 113 | 118
mmol/L | 0.02 (0.44) | -0.06 (0.39) | 0.04 (9.42)

100. Secondary Outcome: Change in Potassium (Week 87)
Description: Change in Potassium was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 112 | 49 | 49
mmol/L | -0.06 (0.45) | 0.00 (0.44) | -0.00 (0.40) | -0.03 (0.43)

101. Secondary Outcome: Change in Sodium (Week 34)
Description: Change in Sodium was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 55 | 108 | 115
mmol/L | 0.1 (2.4) | 0.1 (2.9) | 0.5 (2.7)

102. Secondary Outcome: Change in Sodium (Week 87)
Description: Change in Sodium was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 48 | 49
mmol/L | -0.7 (3.35) | 0.0 (2.92) | -0.3 (2.74) | 0.5 (2.76)

103. Secondary Outcome: Change in Total Protein (Week 34)
Description: Change in total protein was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
g/L | -0.26 (5.48) | -0.97 (4.36) | -0.83 (4.93)

104. Secondary Outcome: Change in Total Protein (Week 87)
Description: Change in total protein was measured from baseline (week -3) until the end of extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
g/L | -1.20 (5.17) | -0.74 (4.88) | -1.31 (4.91) | -1.59 (4.37)

105. Secondary Outcome: Change in Urea (Week 34)
Description: Change in Urea was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
mmol/L | 0.17 (1.27) | -0.40 (1.16) | -0.19 (1.24)

106. Secondary Outcome: Change in Urea (Week 87)
Description: Change in Urea was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
mmol/L | 0.11 (1.40) | -0.21 (1.28) | -0.26 (1.35) | -0.03 (2.46)

107. Secondary Outcome: Change in Uric Acid (Week 34)
Description: Change in Uric acid was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
umol/L | -8.228 (52.557) | -12.61 (50.534) | -21.11 (57.594)

108. Secondary Outcome: Change in Uric Acid (Week 87)
Description: Change in Uric acid was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 112 | 49 | 49
umol/L | -25.22 (59.042) | -21.95 (58.903) | -18.02 (59.716) | -31.31 (86.787)

109. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (GFR) Creatinine (CKD-EPI) (Week 34)
Description: Change in Estimated GFR creatinine (CKD-EPI) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 113 | 118
mL/min/1.73m^2 | -1.34 (10.68) | 2.77 (10.07) | 2.57 (11.24)

110. Secondary Outcome: Change in Estimated GFR Creatinine (CKD-EPI) (Week 87)
Description: Change in estimated GFR creatinine (CKD-EPI) was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 111 | 49 | 49
mL/min/1.73m^2 | 5.36 (12.67) | 2.38 (12.28) | 1.44 (10.52) | 1.67 (15.77)

111. Secondary Outcome: Change in Fasting Plasma Glucose (Week 34)
Description: Change in Fasting plasma glucosewas measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 55 | 112 | 117
mmol/L | 0.01 (0.42) | 0.12 (0.65) | 0.00 (0.56)

112. Secondary Outcome: Change in Fasting Plasma Glucose (Week 87)
Description: Change in Fasting plasma glucose was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 108 | 49 | 48
mmol/L | 0.06 (0.46) | 0.13 (0.77) | 0.05 (0.68) | 0.04 (0.60)

113. Secondary Outcome: Change in Fasting Insulin (Week 34)
Description: Change in Fasting insulin was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 56 | 112 | 117
pmol/L | 14.563 (45.217) | 27.580 (76.230) | 12.778 (53.703)

114. Secondary Outcome: Change in Fasting Insulin (Week 87)
Description: Change in Fasting insulin was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 48 | 48
pmol/L | 12.2 (57.31) | -3.7 (62.39) | -6.5 (53.67) | 13.4 (54.40)

115. Secondary Outcome: Change in Steady State Beta Cell Function (%B) (Week 34)
Description: Change in steady state beta cell function (%B) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of beta cell function
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 53 | 108 | 113
Percentage of beta cell function | 27.10 (105.45) | 36.26 (290.00) | 54.90 (173.14)

116. Secondary Outcome: Change in Steady State Beta Cell Function (%B) (Week 87)
Description: Change in steady state beta cell function (%B) was measured from baseline (week -3) until the end of the week 87.
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of beta cell function
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 105 | 46 | 46
Percentage of beta cell function | 21.72 (154.22) | -16.54 (148.72) | -7.34 (97.62) | 34.54 (161.01)

117. Secondary Outcome: Change in Insulin Resistance (IR %) (Week 34)
Description: Change in Insulin resistance (IR %) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of insulin resistance
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 53 | 109 | 114
Percentage of insulin resistance | 0.53 (1.76) | 1.26 (3.42) | 0.47 (2.32)

118. Secondary Outcome: Change in Insulin Resistance (IR %) (Week 87)
Description: Change in Insulin resistance (IR %) was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of insulin resistance
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 53 | 106 | 46 | 47
Percentage of insulin resistance | 0.50 (2.17) | -0.06 (3.14) | -0.02 (1.99) | 0.52 (2.26)

119. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c) (%) (Week 34)
Description: Change in Glycated haemoglobin (HbA1c) (%) was measured from baseline (week -3) until the end of the main treatment period (week 34).
Time Frame: Week -3, week 34
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | Norditropin | Somapacitan
Number analyzed (Participants) | 57 | 111 | 119
Percentage of HbA1c | 0.04 (0.37) | 0.09 (0.26) | 0.09 (0.31)

120. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c) (%) (Week 87)
Description: Change in Glycated haemoglobin (HbA1c) was measured from baseline (week -3) until the end of the extension treatment period (week 87).
Time Frame: week -3, week 87
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo/Somapacitan | Somapacitan/Somapacitan | Norditropin/Norditropin | Norditropin/Somapacitan
Number analyzed (Participants) | 54 | 110 | 49 | 48
Percentage of HbA1c | 0.09 (0.26) | 0.11 (0.37) | 0.10 (0.28) | 0.07 (0.27)

ADVERSE EVENTS:
Time Frame: Weeks 0-88
Description: All presented AEs are TEAEs. A treatment-emergent AE (TEAE) was defined as an event with onset after first study medicine administration. The results are based on the safety analysis set which included all randomised participants who received at least one dose of trial product.
Groups:
- Placebo - Main Phase: Participants received placebo for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
- Somapacitan - Main Phase: Participants received somapacitan for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
- Norditropin - Main Phase: Participants received Norditropin® for 34 weeks (8 weeks dose titration followed by 26 weeks fixed dose treatment) in the main phase of the trial.
- Somapacitan - Extension Phase: The extension phase treatment period was 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment). This reporting group shows data from the extension phase for the following listed participants: 1) participants who received placebo in the main phase, and switched to receive somapacitan in the extension phase. 2) Participants who received somapacitan in the main phase were continued to receive somapacitan in the extension phase. 3) Participants who received Norditropin® in the main phase and re-randomised at the end of the main phase to receive somapacitan in the extension phase (randomisation was done in a 1:1 manner to receive either somapacitan and Norditropin®).
- Norditropin- Extension Phase: The extension phase treatment period was 52 weeks (8 weeks dose titration followed by 44 weeks fixed dose treatment). This reporting group shows data from the extension phase for the participants who received Norditropin® in the main phase and re-randomised at the end of the main phase to receive Norditropin® in the extension phase (randomisation was done in a 1:1 manner to receive either somapacitan and Norditropin®).
Arm/Group | Placebo - Main Phase | Somapacitan - Main Phase | Norditropin - Main Phase | Somapacitan - Extension Phase | Norditropin- Extension Phase
All-Cause Mortality (participants affected / at risk) | 1/61 | 0/120 | 1/119 | 2/220 | 1/52
Serious Adverse Events (participants affected / at risk) | 5/61 | 7/120 | 12/119 | 15/220 | 3/52
Other Adverse Events (participants affected / at risk) | 29/61 | 53/120 | 55/119 | 85/220 | 27/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Main Phase (N=61) | Somapacitan - Main Phase (N=120) | Norditropin - Main Phase (N=119) | Somapacitan - Extension Phase (N=220) | Norditropin- Extension Phase (N=52)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood testosterone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangiogram (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoconcentration (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Main Phase (N=61) | Somapacitan - Main Phase (N=120) | Norditropin - Main Phase (N=119) | Somapacitan - Extension Phase (N=220) | Norditropin- Extension Phase (N=52)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8) | 11 (11) | 7 (8) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 11 (11) | 4 (4) | 5 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 4 (5) | 5 (5) | 14 (21) | 3 (3)
Fatigue (General disorders) | 2 (2) | 3 (3) | 7 (7) | 9 (11) | 0 (0)
Headache (Nervous system disorders) | 10 (15) | 10 (45) | 11 (50) | 25 (48) | 6 (23)
Hypertension (Vascular disorders) | 1 (1) | 4 (4) | 4 (4) | 3 (3) | 3 (3)
Injection site bruising (General disorders) | 2 (3) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 5 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 9 (12) | 23 (29) | 20 (25) | 33 (41) | 6 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (8) | 5 (14) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 5 (7) | 6 (8) | 7 (17) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 3 (4) | 2 (2) | 3 (4)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 6 (7) | 9 (10) | 17 (18) | 3 (6)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT02229851/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT02229851/SAP_001.pdf